CLINICAL TRIAL: NCT00541580
Title: Comparative Results of Conservatively and Surgically Treated Adolescents With Triplane and Juvenile Tillaux Ankle Fractures After Skeletal Maturity
Status: Terminated | Type: Observational
Sponsor: Hadassah Medical Organization (Other)
Other Study IDs: GOLD-001-HMO-CTIL
Record Dates: First submitted 2007-10-07; First posted 2007-10-10 (Estimated); Last update posted 2011-09-16 (Estimated); Status verified 2011-09

CONDITIONS: Ankle Injuries
MeSH Terms: conditions — Ankle Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Triplane and Juvenile Tillaux fractures of the ankle are well known in adolescent pediatric population. It is widely accepted, that optimal treatment for displaced fractures is close or open reduction and fixation with screws under general anesthesia and under intraoperative fluoroscopy control. Usually a small degree of displacement (up to 2mm) is expected to be healed without any sequences. Until now, no evidence of ankle function and pain after skeletal maturity or long follow-up was published. More than that, no comparative study between operative and no operative treatment of mild and borderline displaced fractures were published.

The purpose of this study is to evaluate functional and radiographic results of operatively and conservatively treated patients after they reach skeletal maturity.

ELIGIBILITY:
Inclusion Criteria:

* Sign informed consent.

Exclusion Criteria:

* Pregnancy
* Unwillingness to sign the informed consent.

Ages: 18 Years to 25 Years | Sex: All
Age Groups: Adult
Study Population: adolescents with triplane and juvenile Tillaux ankle fractures
Sampling Method: Probability Sample

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir Goldman, MD, Principal Investigator — Hadassah Medical Organization; Neum Simanovsky, MD, Study Director — Hadassah Medical Organization; Natalia Simanovski, MD, Study Chair — Hadassah Medical Organization